CLINICAL TRIAL: NCT01765920
Title: Multicentre Double-blind Placebo-controlled Parallel-group Randomized Clinical Trial of Safety and Clinical Efficacy of Ergoferon in Liquid Dosage Form in Treatment of Acute Upper Respiratory Tract Infections in Adult Patients
Brief Title: Clinical Trial of Safety and Efficacy of Ergoferon in Liquid Dosage Form in Treatment of Acute Upper Respiratory Tract Infections in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-ER-006
Record Dates: First submitted 2013-01-09; First posted 2013-01-10 (Estimated); Results first posted 2020-12-11 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-01

CONDITIONS: Acute Upper Respiratory Tract Infections
MeSH Terms: interventions — ergoferon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ergoferon (5 ml 3 times a day) (Experimental): Oral use. Dose per administration: 1 dosing spoon (5ml) without food. For best effect, the solution should be held in the mouth before swallowing.
  Dosing scheme. One dose every 30 minutes for the first 2 hours, followed by three more doses spaced regularly during the rest of the day. From day 2 to 5: 1 spoon taken 3 times daily.
  Interventions: Drug: Ergoferon
- Placebo (5 ml 3 times a day) (Placebo Comparator): Oral use. Placebo using Ergoferon scheme.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ergoferon — 5 ml 3 times a day
  Arms: Ergoferon (5 ml 3 times a day)
Drug: Placebo — 5 ml 3 times a day
  Arms: Placebo (5 ml 3 times a day)

SUMMARY:
The purpose of this study is:

* to evaluate safety of the liquid dosage form of Ergoferon in the treatment of acute upper respiratory tract infections in adults;
* to evaluate clinical efficacy of the liquid dosage form of Ergoferon in the treatment of acute upper respiratory tract infections in adults.

DETAILED DESCRIPTION:
Design: multicenter double-blind placebo-controlled parallel-group randomized clinical trial.

The study will enrol outpatient subjects of either gender aged 18-60 years with clinical manifestations of upper respiratory tract infections (URTI) during seasonal morbidity who are presented to the doctor within the first day of the disease onset. Signed information sheet for the patient is obtained from all participants prior to the screening procedures. Medical history, concomitant medication, tympanic thermometry, patient examination by a doctor, assessment of URTI symptoms severity are performed at screening visit.

URTI symptoms severity examination by the physician is based on Common Cold Questionnaire (CCQ) (PLoS One. 2008; 3(3): e1802. Published online 2008 Mar 19. doi: 10.1371/journal.pone.0001802).

If a patient meets the inclusion criteria and does not have any exclusion criteria, at Visit 1 (Day 1), he/she is randomized into one of two groups: the 1st group (Ergoferon group) patients receive Ergoferon according to the scheme for 5 days; the 2nd group (Placebo group) patients receive placebo according to Ergoferon dosage regimen for 5 days.

The patients are provided with a patient diary where they record tympanic temperature (using tympanic thermometer provided by sponsor) twice a day and URTI symptoms severity according to the Wisconsin Upper Respiratory Symptom Survey - 21 - Daily Symptom Report (WURSS-21©, Wisconsin Upper Respiratory Symptom Survey, 2004.

Created by Bruce Barrett MD PhD et al., UW Department of Family Medicine, 777 S. Mills St. Madison, WI 53715, USA).

In addition, antipyretic administration (if applicable), as well as any possible worsening of the patient's condition (if applicable, for Adverse Events (AEs) evaluation), are also be recorded in a patient diary. An investigator provides the instructions on filling out the diary and helps the patient to make first records of URTI symptoms severity and tympanic temperature in the diary.

Patients are observed up for 7 days (screening and randomization for 1 day, study therapy 1-5 days, the follow-up period for 2 days). During treatment and follow-up period two visits are scheduled (at home or at the study site) on days 3 (Visit 2) and day 7 (Visit 3). At Visits 2 and 3, the investigator will carry out a physical examination, record dynamics of URTI symptoms severity (according to CCQ) and concomitant therapy, and check patient diaries. Treatment compliance is evaluated at Visit 3.

During the study, symptomatic therapy and therapy for underlying chronic conditions are allowed with the exception of the drugs indicated in the section "Prohibited Concomitant Treatment".

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders aged from 18 to 60 years inclusively.
* Patients who visited a doctor during the increase of seasonal incidence within 24 hours after the onset of acute respiratory infection of the upper respiratory tract.
* Body temperature ≥37,8°C at the moment of examination by the doctor.
* Presence of two or more moderate severity symptoms or three or more mild severity symptoms according to the Common Cold Questionnaire (CCQ).
* The possibility to start therapy within 24 hours from the onset of the first symptoms of acute respiratory infection of the upper respiratory tract.
* The use of contraceptive methods by the patients of both the sexes during the study and within 30 days after completion of participation in the study.
* Availability of signed patient information sheet (Informed Consent form) for participation in the clinical trial.

Exclusion Criteria:

* Suspected invasive bacterial infection or the presence of a severe disease requiring use of antibacterial drugs (including sulfanilamides).
* Suspected initial manifestations of diseases that have symptoms similar to acute URTI (other infectious diseases, flu-like symptoms at the onset of systemic connective tissue disorders, hematologic neoplasms and other pathologies).
* Exacerbated or decompensated chronic diseases affecting a patient's ability to participate in the clinical trial.
* Oncological diseases.
* Medical history of polyvalent allergy.
* Allergy/intolerance to any of the components of medications used in the treatment.
* Impaired glucose tolerance, diabetes mellitus type 1 and 2.
* Hereditary fructose intolerance (due to the presence of maltitol in the study drug).
* Use of any medicine listed in the section "Prohibited concomitant treatment" within 30 days preceding the inclusion in this study.
* Pregnancy, breastfeeding.
* Consumption of narcotics, alcohol > 2 alcohol units per day.
* Patients with mental disorders.
* Patients who, from the investigator's point of view, will fail to comply with the observation requirements of the trial or with the regimen of the study drugs.
* Participation in other clinical studies within 3 months prior to enrollment in the current trial.
* Other factors, which hinder the patient's participation in the trial (for example, planned trips or business trips).
* Patients are related to the research staff of the clinical trial site who are directly involved in the trial or are the immediate family member of the researcher. The immediate family members include husband/wife, parents, children or brothers (or sisters), regardless of whether they are natural or adopted.
* Patients employed with MATERIA MEDICA HOLDING (i.e., the company's employee, a part-time employee under contract, or appointed official in charge of the trial, or their immediate family).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 342 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- Russia (18):
  - Non-governmental Health Care Institution "Road Clinical Hospital at the train station Chelyabinsk of OJSC "Russian Railways", Chelyabinsk
  - State Budgetary Educational Institution of Higher Professional Education "Kazan State Medical University", Kazan'
  - Federal State Budgetary Institution "Scientific Research Institute for Vaccines and Serum named after I.I.Mechnikov" of Russian Academy of Medical Science, Moscow
  - State Budgetary Educational Institution of Higher Professional Education "The Russian National Research Medical University named after N.I. Pirogov"/Outpatient Therapy Department of Medicine Faculty, Moscow
  - State Budgetary Educational Institution of Higher Professional Education "The Russian National Research Medical University named after N.I. Pirogov", Moscow
  - Federal State Budgetary Institution "Polyclinic № 3" of Affairs Management Department of the President of Russian Federation, Moscow
  - Municipal Health Care Institution "Podolsk city clinical hospital №3", Podolsk
  - St. Petersburg State Budgetary Health Care Institution " Nevsky Region Сity Polyclinic №25", Saint Petersburg
  - St. Petersburg State Budgetary Health Care Institution "Сity Polyclinic № 117", Saint Petersburg
  - St. Petersburg State Budgetary Health Care Institution "Medical Exercises Dispensary" of Krasnogvardeysky District, Saint Petersburg
  - The Non-governmental Health Care Institution "Road Hospital of the Open Joint Stock Company" Russian Railways", Saint Petersburg
  - State Budgetary Educational Institution of Higher Professional Education "St. Petersburg State Medical University named after I.P. Pavlov", Saint Petersburg
  - Federal State Budgetary Health Care Institution Policlinic № 1 of the Russian Academy of Sciences, Saint Petersburg
  - St. Petersburg State Budgetary Health Care Institution "Сity Polyclinic № 4", Saint Petersburg
  - Regional State Budgetary Health Care Institution "Policlinic № 6", Smolensk
  - State Educational Institution of Higher Professional Education "Voronezh State Medical Academy of N. N. Burdenko" Ministry of Health of the Russian Federation, Voronezh
  - State Budgetary Educational Institution of Higher Professional Education "Yaroslavl State Medical Academy", Yaroslavl
  - State Budgetary Health Care Institution of the Yaroslavl region "Regional Clinical Hospital", Yaroslavl

RESULTS

PARTICIPANT FLOW:
Groups:
- Ergoferon (5 ml 3 Times a Day): Oral use. Dose per administration: 1 dosing spoon (5ml) without food. For best effect, the solution should be held in the mouth before swallowing.
  Dosing scheme. One dose every 30 minutes for the first 2 hours, followed by three more doses spaced regularly during the rest of the day. From day 2 to 5: 1 spoon taken 3 times daily.
  Ergoferon: 5 ml 3 times a day
Period: Overall Study
Arm/Group | Ergoferon (5 ml 3 Times a Day) | Placebo (5 ml 3 Times a Day)
Started | 169 | 173
Completed | 167 | 167
Not Completed | 2 | 6
Not completed — Incorrect inclusion ineligible patient | 2 | 5
Not completed — Patient code disclosure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ergoferon (5 ml 3 Times a Day) | Placebo (5 ml 3 Times a Day) | Total
Number analyzed (Participants) | 169 | 173 | 342
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 169 | 173 | 342
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (10.6) | 35.1 (10.9) | 35.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 115 | 213
  Male | 71 | 58 | 129
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 169 | 173 | 342

OUTCOME MEASURES:

1. Primary Outcome: Average Duration of Fever.
Description: Primary outcome measure is based on the indicators of tympanic thermometry recorded by the patient in the diary during the period of treatment and observation. Thermometry is performed twice a day (morning and evening).
  The criterion of Duration of Fever is the time from enrollment to the first return to the afebrile state or the normalization of tympanic temperature (tympanic temperature ≤37.0 degree Celsius [°C]).
Time Frame: 1-7 days
Population: One patient in the placebo group did not have enough source data for primary outcome analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ergoferon (5 ml 3 Times a Day) | Placebo (5 ml 3 Times a Day)
Number analyzed (Participants) | 167 | 166
days | 3.1 (1.2) | 3.6 (1.4)
Statistical Analysis 1: Comparison: Ergoferon (5 ml 3 Times a Day) vs Placebo (5 ml 3 Times a Day); Test type: Superiority; p = 0.0174, Kruskal-Wallis — A priori threshold for statistical significance α=0.0221 (Pocock boundary for 3 interim analyses)

2. Secondary Outcome: Dynamics of Acute Upper Respiratory Tract Infections (URTI) Symptoms Severity According to the Physical Examination by the Doctor.
Description: Acute URTI symptoms severity is based on the Common Cold Questionnaire (CCQ) and assessed using the "Area under the curve" (AUC) for the total scores on days 1, 3, and 7 of treatment according to the physical examination by the doctor. AUC is calculated by trapezoidal rule. CCQ includes 3 General Symptoms (fevers, chills, muscle pains), 3 Nasal Symptoms (Watery eyes, Runny nose, Sneezing), 1 Throat Symptom (Sore throat), and 2 Chest Symptoms (Cough, Chest pain). Every CCQ symptom is estimated according to the 4-point scoring: none = 0, mild = 1, moderate = 2, severe = 3. Total CCQ scores equal the sum of all scores. The minimum value is 0, and the maximum value is 162. Higher scores mean a worse outcome.
Time Frame: Day 1, 3, and 7.
Population: One patient in the placebo group and one patient in Ergoferon group did not have enough source data for secondary outcome analysis.
Measure: Mean (Standard Deviation); unit: score on a scale*day
Arm/Group | Ergoferon (5 ml 3 Times a Day) | Placebo (5 ml 3 Times a Day)
Number analyzed (Participants) | 166 | 166
score on a scale*day | 25.7 (12.0) | 28.5 (13.9)
Statistical Analysis 1: Comparison: Ergoferon (5 ml 3 Times a Day) vs Placebo (5 ml 3 Times a Day); Test type: Superiority; p = 0.0719, Kruskal-Wallis — A priori threshold for statistical significance α=0.0221 (Pocock boundary for 3 interim analyses)

3. Secondary Outcome: Dynamics of Acute URTI Symptoms Severity According to the Daily Wisconsin Upper Respiratory Symptom Survey - 21 (WURSS-21) Assessment of the Patient (Including the Total WURSS-21 Score, "Symptoms" Domain Score, and "Ability" Domain Score).
Description: Dynamics of symptoms severity according to the WURSS-21 is assessed using the Area under the curve (AUC) for the score for 8 days of the treatment. AUC is calculated by trapezoidal rule. WURSS-21 consists of 21 items (2 questions and 2 domains. Symptoms domain consists of 10 items: Runny nose, Plugged nose, Sneezing, Sore throat, Scratchy throat, Cough, Hoarseness, Head congestion, Chest congestion, Feeling tired. Ability domain consists of 9 items: Think clearly, Sleep well, Breathe easily, Walk, climb stairs, exercise, Accomplish daily activities, Work outside the home, Work inside the home, Interact with others, Live your personal life. The first 20 items are scored according to the 8-point scale (from 0 to 7). The last item is scored according to the 7-point scale: (from 0 to 6). Total WURSS-21 AUC min score=0, max=1169. Symptoms domain min score=0, max=560. Ability domain min score=0, max=504. Higher scores mean a worse outcome.
Time Frame: Days 1 to 8.
Population: One patient in the placebo group did not have enough source data for secondary outcome analysis.
Measure: Mean (Standard Deviation); unit: score on a scale*day
Arm/Group | Ergoferon (5 ml 3 Times a Day) | Placebo (5 ml 3 Times a Day)
Number analyzed (Participants) | 167 | 166
score on a scale*day
  Total WURSS-21 score | 201.6 (106.1) | 236.2 (127.9)
  "Symptoms" domain score | 85.2 (47.6) | 100.4 (54.0)
  "Ability" domain score | 84.3 (58.9) | 102.0 (72.0)
Statistical Analysis 1: Comparison: Ergoferon (5 ml 3 Times a Day) vs Placebo (5 ml 3 Times a Day); Test type: Superiority; p = 0.02, Kruskal-Wallis — Total score analysis. A priori threshold for statistical significance α=0.0221 (Pocock boundary for 3 interim analyses)
Statistical Analysis 2: Comparison: Ergoferon (5 ml 3 Times a Day) vs Placebo (5 ml 3 Times a Day); Test type: Superiority; p = 0.0099, Kruskal-Wallis — "Symptoms" domain analysis. A priori threshold for statistical significance α=0.0221 (Pocock boundary for 3 interim analyses)
Statistical Analysis 3: Comparison: Ergoferon (5 ml 3 Times a Day) vs Placebo (5 ml 3 Times a Day); Test type: Superiority; p = 0.037, Kruskal-Wallis — "Ability" domain analysis. A priori threshold for statistical significance α=0.0221 (Pocock boundary for 3 interim analyses)

4. Secondary Outcome: Percentage of Patients Who Used Antipyretics.
Description: Based on the patient's diary. The outcome is calculated according to the number of patients who were administered the antipyretics due to the fever.
Time Frame: Days 1, 2, 3, 4, and 5.
Population: One patient in the placebo group did not have enough source data for secondary outcome analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Ergoferon (5 ml 3 Times a Day) | Placebo (5 ml 3 Times a Day)
Number analyzed (Participants) | 167 | 166
Participants
  Day 1 | 61 | 72
  Day 2 | 27 | 34
  Day 3 | 7 | 10
  Day 4 | 3 | 4
  Day 5 | 0 | 2
Statistical Analysis 1: Comparison: Ergoferon (5 ml 3 Times a Day) vs Placebo (5 ml 3 Times a Day); Test type: Superiority; p = 0.22, Fisher Exact — Day 1 analysis
Statistical Analysis 2: Comparison: Ergoferon (5 ml 3 Times a Day) vs Placebo (5 ml 3 Times a Day); Test type: Superiority; p = 0.32, Fisher Exact — Day 2 analysis
Statistical Analysis 3: Comparison: Ergoferon (5 ml 3 Times a Day) vs Placebo (5 ml 3 Times a Day); Test type: Superiority; p = 0.47, Fisher Exact — Day 3 analysis
Statistical Analysis 4: Comparison: Ergoferon (5 ml 3 Times a Day) vs Placebo (5 ml 3 Times a Day); Test type: Superiority; p = 0.72, Fisher Exact — Day 4 analysis
Statistical Analysis 5: Comparison: Ergoferon (5 ml 3 Times a Day) vs Placebo (5 ml 3 Times a Day); Test type: Superiority; p = 0.25, Fisher Exact — Day 5 analysis

5. Secondary Outcome: Percentage of Patients Who Have a Worsening of Disease.
Description: The number of patients with the appearance of the lower respiratory tract symptoms, development of complications requiring antibiotics or hospitalization.
Time Frame: Days 1, 2, 3, 4.,5, 6, and 7.
Measure: Count of Participants; unit: Participants
Arm/Group | Ergoferon (5 ml 3 Times a Day) | Placebo (5 ml 3 Times a Day)
Number analyzed (Participants) | 167 | 167
Participants | 3 | 2
Statistical Analysis 1: Comparison: Ergoferon (5 ml 3 Times a Day) vs Placebo (5 ml 3 Times a Day); Test type: Superiority; p = 0.68, Fisher Exact

ADVERSE EVENTS:
Time Frame: 8 days (during the study).
Arm/Group | Ergoferon (5 ml 3 Times a Day) | Placebo (5 ml 3 Times a Day)
All-Cause Mortality (participants affected / at risk) | 0/169 | 0/173
Serious Adverse Events (participants affected / at risk) | 0/169 | 0/173
Other Adverse Events (participants affected / at risk) | 7/169 | 6/173
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ergoferon (5 ml 3 Times a Day) (N=169) | Placebo (5 ml 3 Times a Day) (N=173)
Acute anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increased lymphocytes (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Decreased level of segmented neutrophils (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Increased levels of transaminases (ALT, AST) (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
A large amount of salts in the urine (urates) (Renal and urinary disorders) | 1 (1) | 0 (0)
Increased red blood cells in the urine (Renal and urinary disorders) | 0 (0) | 1 (1)
The presence of mucus in the urine (Renal and urinary disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) — Genyantritis
Acute bilateral rhinosinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Community-acquired pneumonia of the lower lobe of the right lung (Infections and infestations) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Hives
Facial hyperemia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes